CLINICAL TRIAL: NCT00788164
Title: A Phase I Efficacy and Safety Study of HPV16-specific Therapeutic DNA-vaccinia Vaccination in Combination With Topical Imiquimod, in Patients With HPV16+ High Grade Cervical Dysplasia (CIN3)
Brief Title: Vaccine Therapy With or Without Imiquimod in Treating Patients With Grade 3 Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0656; NA_00002176 (Other: JHM IRB); CDR0000617261 (Other: other); 2P50CA098252 (NIH); 1R21CA123876 (NIH)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer; Precancerous Condition; HPV Disease; Human Papilomavirus
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 3; therapeutic vaccine; treatment; CIN; HPV; vaccine; Hopkins; Trimble
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — human papillomavirus vaccine, TA; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Groups 1-3 (Experimental): Patients receive pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine intramuscularly (IM) on days 1 and 29 and TA-HPV vaccine IM on day 57.
  Interventions: Biological: TA-HPV; Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine
- Group 4 (Experimental): Patients receive topical imiquimod on days 1, 29, and 57.
  Interventions: Drug: imiquimod
- Group 5 (Experimental): Patients receive pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine and TA-HPV vaccine as in groups 1-3, and imiquimod as in group 4.
  Interventions: Biological: TA-HPV; Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine; Drug: imiquimod

INTERVENTIONS:
Biological: TA-HPV — Given intramuscularly
  Arms: Group 5; Groups 1-3
Biological: pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine — Given intramuscularly
  Arms: Group 5; Groups 1-3
Drug: imiquimod — Given topically
  Arms: Group 4; Group 5

SUMMARY:
RATIONALE: Vaccines made from DNA or a gene-modified virus may help the body build an effective immune response to kill tumor cells. Biological therapies, such as imiquimod, may stimulate the immune system in different ways and stop tumor cells from growing. Applying topical imiquimod to the cervix may be an effective treatment for cervical intraepithelial neoplasia. Giving vaccine therapy together with imiquimod may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy and to see how well it works when given with or without imiquimod in treating patients with grade 3 cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate safety, tolerability, and feasibility of pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine and TA-HPV vaccine with or without imiquimod in patients with human papillomavirus (HPV)16-positive grade 3 cervical intraepithelial neoplasia (CIN3).

Secondary

* To evaluate the effect of this regimen on histology, based on the regression of cervical intraepithelial neoplasia.
* To evaluate the feasibility and safety of study immunotherapy in these patients.
* To evaluate the quantitative changes in cervical HPV viral load in these patients following study immunotherapy.
* To evaluate changes in lesion size.
* To evaluate the cellular and humoral immune response to vaccination.
* To evaluate local tissue immune response.
* To correlate measures of immune response with clinical response.
* To correlate measures of immune response with those observed in the preclinical model.
* To evaluate if the efficacy of the prime-boost vaccination can be improved with the cervical application of imiquimod.

OUTLINE: This is a dose escalation study of TA-HPV vaccine (groups 1-3 only). Patients are assigned to 1 of 5 treatment groups.

* Groups 1-3: Patients receive pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine intramuscularly (IM) in weeks 0 and 4 and TA-HPV vaccine IM in week 8.
* Group 4: Patients receive topical imiquimod applied to the cervix once in weeks 0, 4, and 8.
* Group 5: Patients receive pNGVL4a-Sig/E7(detox)/HSP70 DNA vaccine and TA-HPV vaccine as in groups 1-3, and imiquimod as in group 4.

Patients experiencing no improvement of their lesions at week 15 undergo standard cone resection of the squamocolumnar junction. If there is either 1) regression of the size of the lesions by colposcopy and/or 2) no CIN3 lesions detected by colposcopy/biopsy and Pap smear and/or 3) significant decrease of HPV viral load, patients are followed until week 28. At that time, loop electrosurgical excision procedure (LEEP) resection is performed if there is a CIN3 lesion detected by colposcopy/biopsy or suspected by Pap smear. Patients undergoing LEEP are followed until week 32. Patients not undergoing LEEP are followed until week 41 to confirm CIN3 regression.

Blood and tissue samples are collected periodically to measure immune response via ELISA, determine viral load and identify co-infecting HPV types via reverse-line blotting, and analyze lymphocytes via flow cytometry.

PROJECTED ACCRUAL: A total of 36 patients (3 in groups 1 and 2, 12 in groups 3 and 5, and 6 in group 4) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Colposcopically and biopsy confirmed grade 3 cervical intraepithelial neoplasia

  * Human papillomavirus (HPV) 16-positive disease by PCR
* Measurable disease after diagnostic biopsy
* No concurrent adenocarcinoma in situ of the cervix

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use an effective form of contraception during study treatment
* Immunocompetent
* No concurrent malignancy, except for nonmelanoma skin lesions
* No serious concurrent disorder, including any of the following:

  * Active systemic infection
  * Autoimmune disease
  * Proven or suspected immunosuppressive disorder
  * Major medical illnesses of the cardiovascular or respiratory system
* No evidence or history of cardiac disease, including any of the following:

  * Congestive heart failure
  * Symptomatic arrhythmia not controlled by medication
  * Unstable angina
  * History of acute myocardial infarction or cerebrovascular accident within the past 6 months
* No history of severe allergy including eczema or other exfoliative skin disorder
* No active eczema within the past 12 months
* No concurrent skin conditions, including any of the following:

  * Burns
  * Traumatic or pruritic skin conditions
  * Open wounds
  * Unhealed surgical scars
* Patients and their close social, sexual, or domestic contacts may not have any of the following active skin diseases:

  * Psoriasis
  * Lichen planus
  * Sever acneiform rash
  * Impetigo
  * Varicella zoster
  * Sepsis
* No close social contact with children under 5 years old
* No close social or domestic contact with a pregnant woman
* No HIV seropositivity
* No allergy to eggs

PRIOR CONCURRENT THERAPY:

* No previous vaccination with vaccinia
* No immunosuppressive medication (i.e., steroid therapy or other immunosuppressive/immunomodulating drugs [e.g., cyclosporine]) within the past 2 months
* No investigational agent(s) within the past 6 months
* No concurrent participation in another experimental protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by number of participants with Serious Adverse Events | 10 weeks from the first intervention
  Presence of Serious Adverse Events (as defined by according to NCI CTCAE v3.0) or dose limiting toxicities related to the study drugs.

SECONDARY OUTCOMES:
Change in histology (CIN3 or no CIN3) of biopsies between baseline and week 15 | 15 weeks from the date of the first intervention
  Absence of CIN3 as assessed by colposcopically directed biopsy at week 15
Change in histology (CIN3 or no CIN3) of biopsies between baseline and week 28 | 28 weeks from the date of the first intervention
  Absence of CIN3 as assessed by colposcopically directed biopsy at week 28.
Quantitative changes in cervical HPV viral load in exfoliated cell samples | 41 weeks from the date of the first intervention
  HPV genotypes present at study entry which become undetectable during the study window
Change in number of lesions by serial digital colposcopy from week 0 to week 15 | Change from baseline to 15 weeks
  Number of lesions that were present at baseline, then become undetectable by colposcopy at week 15
Change in size of lesions by serial digital colposcopy from week 0 to week 15 | Change from baseline to 15 weeks
  Change in size of lesions from baseline to week 15.
Characterization of peripheral and local tissue response to vaccination | 41 weeks
  Compare immune responses in the blood to local immune responses in the tissue for patients who receive the study intervention, from serially obtained peripheral blood specimens and on tissue samples from therapeutic resection
Correlation of immune response with clinical response | 41 weeks
  Compare immune responses in the blood with histologic regression of CIN3 to CIN1 or less
Correlation between measures of immune response and preclinical experimental data | 41 weeks from the date of the first study intervention
  Compare immune responses detected in patients who received the study intervention to those detected in the preclinical animal model.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L. Trimble, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Maldonado L, Teague JE, Morrow MP, Jotova I, Wu TC, Wang C, Desmarais C, Boyer JD, Tycko B, Robins HS, Clark RA, Trimble CL. Intramuscular therapeutic vaccination targeting HPV16 induces T cell responses that localize in mucosal lesions. Sci Transl Med. 2014 Jan 29;6(221):221ra13. doi: 10.1126/scitranslmed.3007323. PMID 24477000
- [Derived] Peng S, Ferrall L, Gaillard S, Wang C, Chi WY, Huang CH, Roden RBS, Wu TC, Chang YN, Hung CF. Development of DNA Vaccine Targeting E6 and E7 Proteins of Human Papillomavirus 16 (HPV16) and HPV18 for Immunotherapy in Combination with Recombinant Vaccinia Boost and PD-1 Antibody. mBio. 2021 Jan 19;12(1):e03224-20. doi: 10.1128/mBio.03224-20. PMID 33468698
- [Derived] Sun YY, Peng S, Han L, Qiu J, Song L, Tsai Y, Yang B, Roden RB, Trimble CL, Hung CF, Wu TC. Local HPV Recombinant Vaccinia Boost Following Priming with an HPV DNA Vaccine Enhances Local HPV-Specific CD8+ T-cell-Mediated Tumor Control in the Genital Tract. Clin Cancer Res. 2016 Feb 1;22(3):657-69. doi: 10.1158/1078-0432.CCR-15-0234. Epub 2015 Sep 29. PMID 26420854
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00788164?term=J0656&recrs=ab&cond=CIN&rank=1